CLINICAL TRIAL: NCT01389557
Title: Evaluation of Impact Dihydroartemisinin-piperaquine Plus Primaquine on Malaria Transmission in Lempasing Village, Lampung Province, Southern Sumatra
Brief Title: Impact of Dihydroartemisinin-piperaquine Plus Primaquine on Malaria Transmission in Lampung Province, Sumatra
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Inge Sutanto, DR Inge Sutanto MPHil, Department of Parasitology, Faculty of Medicine, Indonesia University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 45114-2; 45114 (Other Grant/Funding Number: Bill and Melinda Gates Foundation)
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2011-11

CONDITIONS: Malaria
Keywords: malaria; DHP; PQ; MST
MeSH Terms: conditions — Malaria | interventions — Primaquine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Dihydroartemisinin-piperaquine with primaquine — P. falciparum : Treated with fixed doses of 40 mg dihydroartemisinin and 320 mg piperaquine based on weight for 3 days (D0, D1 and D2) with max dose of 1 x 3 tablets for patients weighing ≥ 41 kg; 1 x 2 tablets for patients weighing 31 - 40 kg, 1 x 1.5 tablets for patients weighing 18 - 30 kg, and 1 X 1 tablet for patients with body weight of 11 - 17 kg. A single dose PQ of 0.75 mg/kg BW was provided on Day-3 using 15 mg base PQ tablets. The maximal dose was 3 tablets for subjects weighing ≥ 60 kg. The dose range for subjects weighing 10 - 13 kg was 0.5 tablet; 14 - 18 kg was 0.75 tablet; 19 - 23 kg was 1 tablet, 24 -30 kg was 1.5 tablet; 31 - 40 kg was 2 tablets; 41- 49 kg was 2.25 tablet; 50 - 59 kg was 2.5 tablet and ≥ 60 kg was 3 tablets.
  P. vivax: DHP (3 days) + primaquine (14 days)
  Other Names: DHP, PQ

SUMMARY:
Artemisinin-based combination therapy (ACT) has been known to be controversial for stopping malaria transmission. The addition of primaquine (PQ) - the only drug commercially available that kills mature transmission stage - to such treatments might be necessary to eliminate this stage. A study is conducted to evaluate the efficacy of dihydroartemisinin-piperaquine (DHP) regimens with PQ on malaria transmission on a community wide level in Lempasing, Lampung, Sumatra.

DETAILED DESCRIPTION:
A mass screening baseline survey enabled the description of malaria prevalence (P. falciparum and P. vivax). Malaria infected asymptomatic (from the mass screening) and symptomatic (malaria infected people attending the health center) people were enrolled in the study. Enrolled malaria infected subjects were treated with DHP and PQ according to the treatment regimen. The community was mass screened for malaria infections every 3 months and an incidence cohort screened every month for infections. The 3 aims were to look at malaria antibodies, haemoglobin levels and the incidence of malaria before and after the drug intervention.

ELIGIBILITY:
Inclusion Criteria:

* All individuals residing Lempasing village, kecamatan Hanura, Lampung province during study period

Exclusion Criteria:

* Individuals with severe or chronic disease (liver, kidney), infant and pregnant or breastfeeding woman
* Individuals that refuse to sign informed consent are excluded.
* normal glucose-6-phosphate dehydrogenase enzyme level based on qualitative test (Trinity Biotech® no 203, USA)
* willingness to sign the informed-consent form

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Presence of malaria (P. falciparum and P. vivax) parasites in blood spot | 6 months
  Finger prick blood samples are collected for malaria blood smear. Thick and thin blood smears were stained with 3% Giemsa solution for 40 minutes and were read under binocular microscope with 1,000X magnification.

CONTACTS AND LOCATIONS:
Overall Officials: Inge Sutanto, Md PhD, Principal Investigator — Univesity of Indonesia
Locations (1):
- Inge Sutanto, Hanura Primary Health Center, Lampung, Sumatra, Indonesia